CLINICAL TRIAL: NCT06577519
Title: Efficacy and Safety of Vicagrel in Patients With With Acute Coronary Syndrome (ACS) Undergoing Percutaneous Coronary Intervention (PCI): a Multi-center, Randomized, Double-blind, Double-dummy , Parallel-controlled, Phase III Trial
Brief Title: Efficacy and Safety Study of Vicagrel in Patients With Acute Coronary Syndrome (ACS) Undergoing Percutaneous Coronary Intervention (PCI)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VCP1-III-01
Record Dates: First submitted 2024-08-28; First posted 2024-08-29 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Acute Coronary Syndrome (ACS) Undergoing Percutaneous Coronary Intervention (PCI)
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — methyl 2-(2-acetoxy-6,7-dihydrothieno(3,2-c)pyridin-5(4H)-yl)-2-(2-chlorophenyl)acetate; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Vicagrel loading followed by Maintenance dose
  Interventions: Drug: Vicagrel
- Control group (Active Comparator): Clopidogrel loading followed by Maintenance dose
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Vicagrel — Vicagrel loading followed by Maintenance dose
  Arms: Experimental group
Drug: Clopidogrel — Clopidogrel loading followed by Maintenance dose
  Arms: Control group

SUMMARY:
This is a multi-center, randomized, double-blind, double-dummy, parallel-controled, phase III trial, aiming to evaluate the effectiveness and safety of long-term continuous administration of Vicagrel capsules in ACS patients undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 80 years old, with no gender restrictions.
* Patients diagnosed with ACS and scheduled for PCI, including STEMI and NSTE-ACS (UA/NSTEMI).
* Voluntarily sign the ICF and be able to follow the visit arrangements specified in the protocol during the trial period.

Exclusion Criteria:

* Expected survival time<12 months;
* Severe liver dysfunction (non heart disease induced ALT or AST>3x ULN) and cirrhosis;
* Pregnant or lactating women, or participants and their partners who plan to become pregnant during the trial period;
* The researchers determined that other reasons were not suitable for participants in this experiment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of MACE | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command of Chinese PLA, Shenyang, Liaoning, China